CLINICAL TRIAL: NCT06986642
Title: Effectiveness of Core Stability Exercises and General Exercises in Patients With Low Back Pain
Brief Title: Core Stability Exercises and General Exercises in Patients With Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REC-01013 Mahroosh
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Low Back Pain
Keywords: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant
Masking Description: this study follows an analytical research model designed effectiveness of core stability exercises and general exercises in patients with low back pain
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Core Stability Exercises
  Interventions: Other: core stability exercises
- Group B (Placebo Comparator): General Exercises
  Interventions: Other: Genreal Exercises

INTERVENTIONS:
Other: core stability exercises — core stability exercises General Exercises
  1. Brisk walking (30 minutes)
  2. Squats (3 sets, 10-15 repetitions)
  3. Lunges (3 sets, 10-15 repetitions per leg)
  4. Push-ups (3 sets, 10-15 repetitions)
  5. Seated row (3 sets, 10-15 repetitions)
  1. Brisk walking (30 minutes) 2. Squats (3 sets, 10-15 repetitions) 3. Lunges (3 sets, 10-15 repetitions per leg) 4. Push-ups (3 sets, 10-15 repetitions) 5. Seated row (3 sets, 10-15 repetitions)
  Arms: Group A
Other: Genreal Exercises — Genreal Exercises
  Arms: Group B

SUMMARY:
Effectiveness of core stability exercises and general exercises in patients with low back pain

DETAILED DESCRIPTION:
The study focuses on understanding core stability exercises and general exercises in patients with low back pain Low back pain (LBP) is an common state with a lifetime occurrence reported to be as high as about 80% . About 5-10% of patients have chronic pain (cLBP), responsible for high direct and indirect (lost production and lost household productivity) costs highly person suffering from disability

ELIGIBILITY:
Inclusion Criteria:

1. Adults (30-45 years)
2. Chronic low back pain (>3 months)
3. Pain intensity ≥ 4/10 on Numeric Pain Rating Scale (NPRS)
4. Ability to perform exercises
5. Willingness to participate and provide informed consent
6. No planned spinal surgery or injection within study duration

Exclusion Criteria:

1. Severe spinal pathology (fracture, tumor, infection)
2. Neurological deficits (numbness, weakness, paralysis)
3. Recent spinal surgery or injection (<6 months)
4. Pregnancy or breastfeeding
5. . Severe mental health conditions (e.g., depression, anxiety)

Musculoskeletal Conditions:

1. Severe osteoporosis
2. Spinal stenosis
3. Scoliosis
4. Recent musculoskeletal injury (<6 months)
5. Fibromyalgia or widespread pain syndr

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-05-13 (Estimated); Study Completion 2026-05-13 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale | 4 weeks
  A numerical rating scale uses numbers to quantify and rank different levels of a characteristic or quality. It's a simple and commonly used tool for assessing subjective experiences like pain or satisfaction. For example, a scale from 1 to 10 could be used to measure pain, with 1 representing no pain and 10 representing the worst imaginable pain

SECONDARY OUTCOMES:
Back pain functional score | 4 weeks
  Stratford et al developed the Back Pain Function Scale (BPFS) to evaluation functional ability in patients with back pain. The authors are from McMaster University Appalachian Physical Therapy (Georgia) and Virginia Commonwealth University.
  1. Brisk walking (30 minutes)
  2. Squats (3 sets, 10-15 repetitions)
  3. Lunges (3 sets, 10-15 repetitions per leg)
  4. Push-ups (3 sets, 10-15 repetitions)
  5. Seated row (3 sets, 10-15 repetitions)

CONTACTS AND LOCATIONS:
Overall Officials: Ataur Rahman, MS-PT (CPPT), Principal Investigator — Riphah International University
Locations (1):
- Riphah international University malakand campus, Malakand, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No